CLINICAL TRIAL: NCT04259060
Title: Hydroxocobalamin Approach for Reducing of Calprotectin With Butyrate for Ulcerative
Brief Title: Hydroxocobalamin Approach for Reducing of Calprotectin With Butyrate for Ulcerative Colitis Remission
Acronym: HARBOUR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to pursue a smaller scale pilot study instead
Sponsor: Joshua Korzenik (Other)
Responsible Party: Sponsor-Investigator, Joshua Korzenik, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P003412
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Butyrate; Hydroxocobalamin
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Hydroxocobalamin; Butyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxocobalamin with Butyrate (Active Comparator): Subjects enrolled will take hydroxocobalamin capsules twice daily for 4 weeks. All subjects will take an oral butyrate dose of 120 mg twice daily for 4 weeks.
  Interventions: Drug: Hydroxocobalamin with Butyrate
- Placebo with Butyrate (Placebo Comparator): Subjects enrolled will take placebo capsules twice daily for 4 weeks. All subjects will take an oral butyrate dose of 120 mg twice daily for 4 weeks.
  Interventions: Drug: Placebo with Butyrate

INTERVENTIONS:
Drug: Hydroxocobalamin with Butyrate — In phase 1, patients will take hydroxocobalamin at 1g daily for four weeks. This will be in the form of 1 500mg capsule twice a day. Butyrate will be 240 mg daily in a divided dose (120 mg twice daily) which is 5 pills twice a day.
  In phase 2, the dose of hydroxocobalamin will be increased to 2g daily (1g twice a day) for four weeks pending FDA approval. Butyrate will remain at 240 mg daily in a divided dose (120 mg twice daily) which is 5 pills twice a day. Patients will undergo flexible sigmoidoscopy at baseline and at week four in phase 2.
  Arms: Hydroxocobalamin with Butyrate
Drug: Placebo with Butyrate — In phase 1, patients will take 1 placebo capsule twice a day. Butyrate will be taken at 240 mg daily in a divided dose (120 mg twice daily) which is 5 pills twice a day.
  In phase 2, patients will take 2 placebo capsules twice a day, along with butyrate at 240 mg daily in a divided dose (120 mg twice daily) which is 5 pills twice a day.
  Arms: Placebo with Butyrate

SUMMARY:
This is a 4-week pilot, multicenter, randomized, double-blinded placebo controlled trial of hydroxocobalamin and butyrate in ulcerative colitis (UC) that will occur in two phases. The main objectives of this study are to determine the capacity of hydroxocobalamin and butyrate to reduce calprotectin in those with inflammatory disease in UC to determine the safety and preferential dose of hydroxocobalamin with butyrate in UC.

DETAILED DESCRIPTION:
The goal of this study is to determine the preferable dose of hydroxocobalamin in a 4-week pilot study in patients with UC and determine if this approach can reduce stool calprotectin. Before going forward with a larger efficacy trial, the investigators are first aiming to determine if the supplements/medications we are proposing to use are sufficient to reduce a biomarker. Consequently, this study will look at a more easily measurable biomarker to provide evidence that the dosing is sufficient.

This pilot study will be conducted to assess preferable dose of hydroxocobalamin based on reduction of calprotectin. The investigators aim to determine if this reduction is sustained over time and is correlated to changes in clinical disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Ability to give consent
3. Patients with a confirmed diagnosis of UC for > 3 months
4. History of > 15 cm of colonic involvement as confirmed by colonoscopy
5. Disease activity based on calprotectin > 200
6. Allowed medications: mesalamine and sulfasalazine
7. Partial Mayo score of > 4 for phase one or a total Mayo score > 5 in phase 2
8. Patients with primary sclerosing cholangitis are eligible to enroll

Exclusion Criteria:

1. History of uncontrolled hypertension with a systolic BP > 140 and a systolic BP > 90
2. Chronic kidney disease as defined by a GFR <60mL/min
3. Impaired hepatic function (transaminases elevated > 2.5 x ULN) unless due to PSC
4. Evidence of C. difficile - negative test result within 1 month is acceptable to confirm
5. Infectious Colitis or drug induced colitis
6. Crohn's Disease or Indeterminate colitis
7. Decompensated liver disease
8. Patients who are pregnant or breastfeeding
9. Prohibited medications: Vitamin C, prednisone, immune modulators (including but not limited to azathioprine, 6-mercaptopurine, mycophenolate mofetil, tacrolimus, cyclosporine, thalidomide, interleukin-10 and interleukin-11) and anti-TNF agents within the past six weeks
10. Use of rectal therapies
11. Patients who have a confirmed malignancy or cancer within 5 years
12. Participation in a therapeutic clinical trial in the preceding 30 days or simultaneously during this trial
13. Congenital or acquired immunodeficiencies
14. Other comorbidities including: Diabetes mellitus, systemic lupus
15. Patients with a history of kidney stones
16. Patients with a history or risk of cardiovascular conditions, including arrhythmia, long QT syndrome, congestive heart failure, stroke, or coronary artery disease
17. High likelihood of colectomy in the next 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline fecal calprotectin at week 4 | At baseline and at week 4
  Proportion of patients with reductions in fecal calprotectin
Incidence of Treatment-Emergent Adverse Events (AE) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) | Up to 4 weeks
  CTCAE are a set of criteria for the standardized classification of adverse effects of drugs used in clinical trials. It uses a range of grades from 1 to 5, where 1 is mild and 5 is life-threatening.The number of AE and grade of each AE will be measured for the duration of the trial.
Clinical Symptoms assessed by Simple Clinical Colitis Activity Index (SCCAI) | Up to 4 weeks
  The SCCAI is an index to measure disease activity in patients with UC. SCCAI will be used throughout the trial to measure clinical UC symptoms of participants.

SECONDARY OUTCOMES:
Assessment of urinary and plasma nitrite, nitrate levels and nitrosothiol levels | At week 1-2 and at week 4
  Comparison of levels at baseline to week 1-2 and week 4
Normalization of fecal calprotectin below the upper limit of normal | At the end of week 4
  Assessment in number of patients whose fecal calprotectin normalizes
Reduction of Mayo Score (Phase 2) | At the end of week 4
  Proportion of patients with a reduction in Mayo Score
Correlation between urinary and plasma nitrite, nitrate or nitrosothiol levels and fecal calprotectin | Up to 4 weeks
  Comparison of biochemical levels with calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Korzenik, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No